CLINICAL TRIAL: NCT02832622
Title: MultiPoint Pacing™ Post Market Study
Acronym: MPP-PMS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10149
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
Keywords: MultiPoint Pacing; Heart Failure; Cardiac Resynchronization Therapy; SJM Quadripolar Biventricular Pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MPP Programming: This post-market study was designed to characterize the real-world use of MPP technology in patients indicated for CRT device implant. Therefore in order to adequately characterize MPP, data from subjects with MPP programmed continuously or for at least 3 months prior to the final follow-up are reported as the MPP programming group.
  Interventions: Device: MPP; Device: BiV/MPP

INTERVENTIONS:
Device: MPP — MPP ON within 1 month post implant and then continuously programmed ON until 12 months (i.e., MPP ON for months 1-12 continuously)
Device: BiV/MPP — MPP ON at the 12-month study visit and for at least 3 continuous months prior to 12-month assessment (i.e., BiV pacing ON at some point in months 1-9 and MPP ON for months 10-12)

SUMMARY:
This is a prospective, multicenter, non-randomized registry/observational study. The study will enroll up to 2,000 patients with successful St. Jude Medical (SJM) Cardiac Resynchronization Therapy (CRT) MP device implant from up to 140 centers undergoing CRT implantation.

DETAILED DESCRIPTION:
Any patient who received a market approved SJM Quadra Allure MP, Quadra Assura MP, or newer SJM CRT MP device is eligible for enrollment in the study. MultiPoint Pacing (MPP) programming guidance will be specified in the protocol. Patients will be followed for 12 months after implant. Data will be collected at Baseline (within 30 days prior to implant), Post-Implant (within 30 days following successful CRT device implant), 3, 6, 12 months and during any unscheduled follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled to receive a new CRT implant or an upgrade from an existing implantable cardioverter defibrillator or pacemaker implant (SJM CRT MP device and SJM Quadripolar Lead) with no prior left ventricular lead placement
* Have the ability to provide informed consent for study participation and are willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Are expected to receive a heart transplant during the duration of the study
* Have an epicardial ventricular lead system (Active or Inactive)
* Are less than 18 years of age
* Are currently participating in a clinical investigation including an active treatment arm and belong to the active arm
* Are not expected to complete the study follow-up schedule or duration due to any health condition other than heart failure, such as malignancy, indication for heart transplant or hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are indiciated for a Cardiac Resynchronization Therapy (CRT) device
Sampling Method: Probability Sample
Enrollment: 2169 (Actual)
Dates: Start 2016-07; Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay Cohorn, Study Director — Abbott Medical Devices
Locations (128):
- United States (110):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Heart Center Research, LLC., Huntsville, Alabama
  - Integrated Medical Services, Avondale, Arizona
  - Cardiovascular Consultants Ltd, Glendale, Arizona
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - John C. Lincoln North Mountain Hospital, Phoenix, Arizona
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Comprehensive Cardiovascular Specialists, Alhambra, California
  - USC University Hospital, Los Angeles, California
  - Jeffrey Goodman, Los Angeles, California
  - Premier Cardiology, Inc, Newport Beach, California
  - Desert Heart Rhythm Consultants, Palm Springs, California
  - Chaparral Medical Group, Pomona, California
  - Cardiac Rhythm Specialists, Inc., Reseda, California
  - San Diego Cardiac Center, San Diego, California
  - COR Healthcare Medical Associates, Torrance, California
  - Aurora Denver Cardiology Associates, P.C., Aurora, Colorado
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - Cardiac Arrhythmia Services, Boca Raton, Florida
  - Yoel R. Vivas, MD, Delray Beach, Florida
  - Heart Rhythm Solutions, Hollywood, Florida
  - Citrus Cardiology Consultants, PA, Inverness, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Naushad Shaik, MD, Kissimmee, Florida
  - Jorge Diaz, M.D., P.A., Lake Mary, Florida
  - Central Florida Medical Research, New Smyrna Beach, Florida
  - Usman R. Siddiqui, MD, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Brevard Cardiovascular Research Associates, Inc., Rockledge, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - VA Medical Center - Tampa, Tampa, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Coliseum Medical Centers, Macon, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Illinois Heart and Vascular - Hinsdale, Hinsdale, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Reid Health, Richmond, Indiana
  - Healient Physician Group, Leawood, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - One Health Cardiology, Owensboro, Kentucky
  - Gregory C. Sampognaro Interventional Cardiology, Monroe, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Trinity Health-Michigan d/b/a Michigan Heart, Ann Arbor, Michigan
  - Michigan Electrophysiology Specialists, Flushing, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - MidMichigan Medical Center-Midland, Midland, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - St. Louis Heart and Vascular PC, St Louis, Missouri
  - Kearney Regional Medical Center, Kearney, Nebraska
  - BryanLGH Medical Center East, Lincoln, Nebraska
  - HealthCare Partners Cardiology, Las Vegas, Nevada
  - Catholic Medical Center, Manchester, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Atlantic Health System - Morristown Memorial Hospital, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - St. Peter's Health Partners Medical Associates, PC, Albany, New York
  - Trinity Medical WNY, PC, Buffalo, New York
  - Novant Health Heart and Vascular Research Institute, Charlotte, North Carolina
  - VA Medical Center Durham, Durham, North Carolina
  - Highpoint Regional Hospital, High Point, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals Elyria Medical Center, Elyria, Ohio
  - Middletown Cardiovascular Associates, Middletown, Ohio
  - Samaritan Heart & Vascular Institute - Cardiology Dept., Corvallis, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Presbyterian Medical Center (PA), Philadelphia, Pennsylvania
  - Scranton Cardiovascular Physicians, Scranton, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Pee Dee Cardiology Associates, PA, Florence, South Carolina
  - St. Francis Hospital, Greenville, South Carolina
  - Lexington Cardiology, Lexington, South Carolina
  - Mountain States Medical Group Cardiology, Johnson City, Tennessee
  - Cardiovascular Associates, PC (Wellmont Holston Valley M C), Kingsport, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Austin Heart, Austin, Texas
  - HeartPlace, Bedford, Texas
  - Fort Worth Heart, Fort Worth, Texas
  - Houston Cardiovascular Associates, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Cardiology Clinic Of San Antonio Pa, San Antonio, Texas
  - Wichita Falls Heart Clinic, Wichita Falls, Texas
  - McKay-Dee Heart Services, Ogden, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Heart - The Cardiovascular Group, P.C., Falls Church, Virginia
  - Bayview Physicians Services, PC, Virginia Beach, Virginia
  - Kootenai Heart Clinics, Spokane, Washington
  - St. Mary's Hospital, Huntington, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
  - Wheaton Franciscan Medical Group - Heart Rhythm Specialists, Wauwatosa, Wisconsin
- Argentina (3):
  - Instituto Argentino de Diagnostico y Tratamiento, Caba, Buenos Aires
  - Fundacion Favaloro para la Docencia e Inv. med., Buenos Aires, Rio de La Plata
  - Instituto Cardiovascular Buenos Aires (ICBA), Buenos Aires, Rio de La Plata
- Colombia (2):
  - Fundacion Clinica Shaio, Bogota, Antioquia
  - APEX Foundation, Medellín, Antioquia
- Japan (13):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Akashi Medical Center, Hyōgo, Kinki
  - Tohoku University Hospital, Sendai, Miyagi
  - Tokyo Women's Medical University, Shinjuku-Ku, Tokyo
  - Chiba University, Chiba
  - St. Marianna University School of Medicine Hospital, Kanagawa
  - Shinshu University Hospital, Matsumoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Sakurabashi Watanabe Hospital, Osaka
  - National Cerebral and Cardiovascular Center Hospital, Osaka
  - Osaka University Hospital, Osaka
  - University of Tsukuba Hospital, Tsukuba

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This post-market study was designed to characterize the real-world use of MPP technology in patients indicated for CRT device implant. Therefore in order to adequately characterize MPP, data from subjects with MPP programmed continuously or for at least 3 months prior to the final follow-up are reported as the MPP programming group and the associated results presented.
Groups:
- MPP Programming: Data from subjects with MPP programmed continuously or for at least 3 months prior to the final follow-up are reported as the MPP programming group.
Period: Overall Study
Arm/Group | MPP Programming
Started | 2169
Completed (Sixteen (16) cardiovascular deaths were included in the 433 subjects who completed the trial as they met one of the endpoint of the trial.) | 433
Not Completed | 1736
Not completed — MPP not programmed | 1259
Not completed — Withdrawal by Subject | 123
Not completed — Death | 119
Not completed — Unsuccessful CRT implant | 93
Not completed — Lost to Follow-up | 45
Not completed — Patient non-compliance | 42
Not completed — Withdrawal by other reasons | 25
Not completed — System explant | 24
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Population: Subjects programmed with MPP are included in the analysis population
Groups:
- MPP Group: MPP Group: Subjects programmed with MPP in the study are included in the analysis population.
Arm/Group | MPP Group
Number analyzed (Participants) | 433
Age, Continuous [Mean (Standard Deviation); unit: Age] | 70.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 316
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 338
  Black or African American | 35
  Asian | 19
  Hispanic or Latino | 34
  Other | 7
Region of Enrollment [Number; unit: participants]
  Colombia | 3
  Argentina | 4
  United States | 414
  Japan | 12
Quality of Life (MLWHF) [Mean (Standard Deviation); unit: scores on a scale] — MLWHF score: the total scale is from 0 to 105, with higher scores indicating worse health status. Population: A baseline population differs from the overall due to missing data points.
  scores on a scale
    number analyzed (Participants) | 430
    (all) | 39.9 (28.1)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percentage] — Population: A baseline population differs from the overall due to missing data points.
  Percentage
    number analyzed (Participants) | 386
    (all) | 29.7 (10.4)
Left Ventricular End-Systolic Volume [Mean (Standard Deviation); unit: mL] — Population: A baseline population differs from the overall due to missing data points.
  mL
    number analyzed (Participants) | 123
    (all) | 113.9 (67.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of CRT Responders as Measured by the Clinical Composite Score (CCS)
Description: The CCS has 4 components: New York Heart Association (NYHA) functional classification, Patient Global Assessment (PGA), heart failure (HF) events, cardiovascular death. NYHA Class ranges from Class I (least severe) to Class IV (most severe); possible PGA responses are "markedly worse", "moderately worse", "slightly worse", "no change", "slightly better", "moderately better, "markedly better". CCS components were used to classify or score subjects as "IMPROVED" (at least one-class improvement in NYHA Class or improvement by PGA "moderately" or "markedly" better AND no HF events AND no cardiovascular death), or "WORSENED" (worsening in NYHA Class OR worsening by PGA "moderately" or "markedly" worse OR presence of HF events OR Cardiovascular death, or "UNCHANGED" (neither "improved" or "worsened"). Note CCS is not a numeric score. A responder is defined as improved or unchanged from baseline and non-responder is defined as worsened from baseline.
Time Frame: One year
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Count of Participants; unit: Participants
Groups:
- MPP Group: Subjects programmed with MPP in the study are included in the analysis population.
Arm/Group | MPP Group
Number analyzed (Participants) | 433
Participants | 350

2. Other Pre Specified Outcome: Change in Quality of Life
Description: The change in the Minnesota Living with Heart Failure (MLWHF) questionnaire score between baseline and 12 months (12 months - baseline).
  MLWHF score: the total scale is from 0 to 105, with higher scores indicating worse health status.
Time Frame: baseline and one year
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MPP Group
Number analyzed (Participants) | 406
score on a scale | -17.4 (24.4)

3. Other Pre Specified Outcome: Duration of MPP Programming in Months
Description: The duration of MPP programming in months in the treatment groups.
Time Frame: One year
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | MPP Group
Number analyzed (Participants) | 433
Months | 10.43 (2.58)

4. Other Pre Specified Outcome: Number of MPP Programming Optimizations Per Subject
Description: The number of MPP programming optimizations per subject
Time Frame: One year
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Mean (Standard Deviation); unit: programming optimizations
Arm/Group | MPP Group
Number analyzed (Participants) | 433
programming optimizations | 0.73 (0.74)

5. Other Pre Specified Outcome: Number of Subjects With Heart Failure Hospitalization
Description: HF event is defined as any one of the following when the subject has symptoms and/or signs consistent with congestive heart failure:
  * Hospitalization for HF ≥ 24 hours
  * Clinic or hospital visit for HF<24 hours (i.e. outpatient treatment, observational care, ER, Urgent Care and physician's office visit) requiring administration of IV diuretics, inotropes, and/or vasodilators
Time Frame: One year
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Count of Participants; unit: Participants
Arm/Group | MPP Group
Number analyzed (Participants) | 433
Participants | 57

6. Other Pre Specified Outcome: Number of Subjects With Cardiovascular Hospitalization
Description: Number of subjects with cardiovascular hospitalization as reported by the sites
Time Frame: One year
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Count of Participants; unit: Participants
Arm/Group | MPP Group
Number analyzed (Participants) | 433
Participants | 142

7. Other Pre Specified Outcome: Number of Subjects With Heart Failure 30-day Hospitalization
Description: Number of subjects with heart failure 30-day hospitalization as reported by the sites
Time Frame: 30 days
Population: The analysis population includes any subjects whose device is programmed with MPP.
Measure: Count of Participants; unit: Participants
Arm/Group | MPP Group
Number analyzed (Participants) | 433
Participants | 6

8. Other Pre Specified Outcome: Number of Deaths
Description: Overall mortality rate for all subjects who started the trial is summarized.
Time Frame: One year
Population: The analysis population includes any subjects who started the trial.
Measure: Count of Participants; unit: Participants
Groups:
- MPP Programming: Overall mortality rate for all subjects who started the trial is summarized.
Arm/Group | MPP Programming
Number analyzed (Participants) | 2169
Participants | 135

9. Other Pre Specified Outcome: Change in Left Ventricular Ejection Fraction
Description: Change in left ventricular ejection fraction between baseline and 12 months (12 months - baseline)
Time Frame: baseline and one year
Population: The analysis population includes any subjects whose device is programmed with MPP. LVEF was optional data point in the study. Results were available from a very small number of subjects.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | MPP Group
Number analyzed (Participants) | 81
percentage | 11.9 (12.0)

10. Other Pre Specified Outcome: Change in Left Ventricular End Systolic Volume
Description: Change in left ventricular end systolic volume between baseline and 12 months (Baseline - 12 months)
Time Frame: baseline and one year
Population: The analysis population includes any subjects whose device is programmed with MPP. LVESV was optional data point in the study. Results were available from a very small number of subjects.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MPP Group
Number analyzed (Participants) | 20
mL | 22.5 (57.3)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Overall Study Cohort: All patients who started in the study are included in the all-cause mortality, serious adverse events and/or other adverse events tables.
Arm/Group | Overall Study Cohort
All-Cause Mortality (participants affected / at risk) | 135/2169
Serious Adverse Events (participants affected / at risk) | 821/2169
Other Adverse Events (participants affected / at risk) | 288/2169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Cohort (N=2169)
Abnormal Labs (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Angina (Cardiac disorders) | 2 (2)
Aortic Insufficiency (Cardiac disorders) | 1 (1)
Aortic Stenosis (Cardiac disorders) | 1 (1)
Atherosclerotic Cardiovascular Disease (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 12 (12)
Cardiac Arrhythmias (Cardiac disorders) | 72 (80)
Cardiac Sarcoidosis (Cardiac disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 6 (6)
Carotid Stenosis (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 10 (10)
Dilated Cardiomyopathy (Cardiac disorders) | 3 (3)
Heart Failure Exacerbation (Cardiac disorders) | 168 (227)
Hypotension (Cardiac disorders) | 5 (5)
Hypotensive Shock (Cardiac disorders) | 1 (1)
Lightheadedness (Cardiac disorders) | 1 (1)
Loss Of Capture (Cardiac disorders) | 1 (1)
Mitral Regurgitation (Cardiac disorders) | 1 (1)
Multi-Organ Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Non-St-Elevation Myocardial Infarction (Cardiac disorders) | 12 (14)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pulmonary Edema (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 2 (2)
Valve Damage (Cardiac disorders) | 2 (2)
Heart Failure Exacerbation (Ear and labyrinth disorders) | 1 (1)
Abnormal Labs (Endocrine disorders) | 1 (1)
Diabetes (General disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Excessive Bleeding (Gastrointestinal disorders) | 4 (4)
Gallstone (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 12 (12)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Peritonits (Gastrointestinal disorders) | 1 (1)
Abnormal Labs (General disorders) | 2 (2)
Accidental Injury (General disorders) | 2 (2)
Allergic Reaction (General disorders) | 2 (3)
Altered Mental Status (General disorders) | 4 (4)
Anemia (General disorders) | 7 (7)
Ascites (General disorders) | 1 (1)
Cardiac Arrest (General disorders) | 7 (7)
Cardiac Arrhythmias (General disorders) | 4 (4)
Cardio-Respiratory Failure (General disorders) | 1 (1)
Chest Pain (General disorders) | 13 (13)
Confusion (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Dehydration (General disorders) | 2 (2)
Device Discharge (General disorders) | 1 (1)
Diarrhea (General disorders) | 1 (1)
Drug Toxicity (General disorders) | 2 (2)
Dyspnea (General disorders) | 4 (5)
Encephalopathy (General disorders) | 3 (3)
Excessive Bleeding (General disorders) | 2 (2)
Gastrointestinal Bleeding (General disorders) | 1 (1)
Heart Failure Exacerbation (General disorders) | 5 (5)
Hematoma/Seroma (General disorders) | 3 (3)
Hepato-Renal Failure (General disorders) | 1 (1)
Hernia (General disorders) | 2 (2)
Hypertension (General disorders) | 1 (1)
Hypotension (General disorders) | 6 (6)
Hypoxia (General disorders) | 2 (2)
Medication Error (General disorders) | 1 (1)
Metabolic Bone Disease (General disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 3 (3)
Myocardial Infarction (General disorders) | 1 (1)
Nausea and Vomiting (General disorders) | 1 (1)
Non-Cardiac Death (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pericardial Effusion (General disorders) | 2 (2)
Pleural Effusion (General disorders) | 5 (5)
Pre-Syncope (General disorders) | 1 (1)
Pulmonary Edema (General disorders) | 6 (6)
Renal Failure (General disorders) | 4 (4)
Respiratory Failure (General disorders) | 9 (9)
Rhabdomyolysis (General disorders) | 1 (1)
Sepsis (General disorders) | 1 (1)
Syncope (General disorders) | 6 (6)
Twiddler's Syndrome (General disorders) | 1 (1)
Unresponsiveness (General disorders) | 1 (1)
Weakness (General disorders) | 2 (2)
Acute Hepatitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cirrhosis (Hepatobiliary disorders) | 1 (1)
Dyspnea (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 80 (90)
Pneumonia (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 11 (11)
Septic Shock (Infections and infestations) | 1 (1)
Accidental Injury (Injury, poisoning and procedural complications) | 18 (18)
Cardiac Arrhythmias (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 5 (5)
Cardiac/Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 1 (1)
Cardiac/Coronary Sinus Perforation (Injury, poisoning and procedural complications) | 4 (4)
Deep Vein Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Drug Overdose (Injury, poisoning and procedural complications) | 1 (1)
Excessive Bleeding (Injury, poisoning and procedural complications) | 2 (2)
Hematoma/Seroma (Injury, poisoning and procedural complications) | 12 (12)
Infection (Injury, poisoning and procedural complications) | 3 (3)
Pain (Injury, poisoning and procedural complications) | 1 (1)
Pericarditis (Injury, poisoning and procedural complications) | 1 (1)
Pneumothorax/Hemothorax (Injury, poisoning and procedural complications) | 7 (7)
Pulmonary Edema (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Renal Failure From Contrast Media Used To Visualize Coronary Veins (Injury, poisoning and procedural complications) | 1 (1)
Thrombolytic or Air Embolism (Injury, poisoning and procedural complications) | 2 (2)
Wound Site Complications (Injury, poisoning and procedural complications) | 2 (2)
Abnormal Labs (Investigations) | 3 (3)
Chest Pain (Investigations) | 1 (1)
Drug Toxicity (Investigations) | 1 (1)
Induced Atrial or Ventricular Arrhythmias (Investigations) | 1 (1)
Rise in Threshold and Exit Block (Investigations) | 1 (1)
Accidental Injury (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Colon Polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14)
Cerebellar Hemorrhage (Nervous system disorders) | 2 (2)
Cerebral Hemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2)
Glioblastoma (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 3 (3)
Cardiac Arrhythmias (Product Issues) | 1 (1)
Cardiac/Coronary Sinus Perforation (Product Issues) | 1 (1)
Change in Thresholds (Product Issues) | 3 (3)
Device Malfunction (Product Issues) | 1 (1)
Elevated Defibrillation Threshold (Product Issues) | 1 (1)
Induced Atrial or Ventricular Arrhythmias (Product Issues) | 1 (1)
Infection (Product Issues) | 1 (1)
Lead Dislodgement (Product Issues) | 35 (38)
Lead/Port Damage (Product Issues) | 1 (1)
Loss of Capture (Product Issues) | 2 (2)
Loss of Pacing and/or Sensing due to Dislodgement or Mechanical Malfunction of The Pacing Lead (Product Issues) | 5 (5)
Oversensing (Product Issues) | 1 (1)
Pectoral/Diaphragmatic/Phrenic Nerve Stimulation (Product Issues) | 1 (1)
Rise in Threshold And Exit Block (Product Issues) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cholecystitis (Renal and urinary disorders) | 1 (1)
Dialysis Shunt Occlusion (Renal and urinary disorders) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 4 (4)
Renal Failure (Renal and urinary disorders) | 20 (23)
Renal Transplantation (Renal and urinary disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Accidental Injury (Social circumstances) | 1 (1)
Wound Site Complications (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 3 (3)
AV Fistula (Vascular disorders) | 1 (1)
Carotid Stenosis (Vascular disorders) | 2 (2)
Cerebrovascular Accident (Vascular disorders) | 4 (4)
Deep Vein Thrombosis (Vascular disorders) | 3 (3)
Excessive Bleeding (Vascular disorders) | 1 (1)
Limb Ischemia (Vascular disorders) | 1 (1)
Occluded Stent (Vascular disorders) | 1 (1)
Peripheral Artery Disease (Vascular disorders) | 1 (1)
Peripheral Vascular Disease (Vascular disorders) | 1 (1)
Ruptured Abdominal Aortic Aneurysm (Vascular disorders) | 1 (1)
Stroke (Vascular disorders) | 6 (6)
Thrombolytic or Air Embolism (Vascular disorders) | 3 (3)
Transient Ischemic Attack (Vascular disorders) | 1 (1)
Ulcer (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Cohort (N=2169)
Thrombolytic or Air Embolism (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrhythmias (Cardiac disorders) | 7 (7)
Dyspnea (Cardiac disorders) | 1 (1)
Heart Failure Exacerbation (Cardiac disorders) | 4 (4)
Lead Dislodgement (General disorders) | 3 (3)
Pectoral/Diaphragmatic/Phrenic Nerve Stimulation (General disorders) | 9 (9)
Allergic Reaction (General disorders) | 3 (3)
Altered Mental Status (General disorders) | 1 (1)
Change in Thresholds (General disorders) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Device Vibration (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dyspnea (General disorders) | 1 (1)
Hematoma/Seroma (General disorders) | 3 (3)
Hypertension (General disorders) | 1 (1)
Hypotension (General disorders) | 2 (2)
Lead Dislodgement (General disorders) | 1 (1)
Loss of Capture (General disorders) | 2 (2)
Pain (General disorders) | 4 (4)
Loss Of CapturePectoral/Diaphragmatic/Phrenic Nerve Stimulation (General disorders) | 7 (8)
Pre-Syncope (General disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Accidental Injury (Injury, poisoning and procedural complications) | 2 (2)
Anemia (Injury, poisoning and procedural complications) | 2 (2)
Cardiac/Coronary Sinus Dissection (Injury, poisoning and procedural complications) | 5 (5)
Deep Vein Thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Excessive Bleeding (Injury, poisoning and procedural complications) | 3 (3)
Hematoma/Seroma (Injury, poisoning and procedural complications) | 13 (13)
Infection (Injury, poisoning and procedural complications) | 1 (1)
Pain (Injury, poisoning and procedural complications) | 3 (3)
Pericardial Effusion (Injury, poisoning and procedural complications) | 2 (2)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Thrombolytic or Air Embolism (Injury, poisoning and procedural complications) | 1 (1)
Transient Ischemic Attack (Injury, poisoning and procedural complications) | 1 (1)
Wound Site Complications (Injury, poisoning and procedural complications) | 3 (3)
Increased Impedance (Investigations) | 1 (1)
Induced Atrial or Ventricular Arrhythmias (Investigations) | 1 (1)
Change in Thresholds (Product Issues) | 22 (23)
Device Discharge (Product Issues) | 1 (1)
Inappropriate Therapy (Product Issues) | 2 (2)
Induced Atrial or Ventricular Arrhythmias (Product Issues) | 1 (1)
Lead Dislodgement (Product Issues) | 32 (32)
Lead/Port Damage (Product Issues) | 1 (1)
Loss of Capture (Product Issues) | 12 (12)
Loss of Pacing and/or Sensing due to Dislodgement or Mechanical Malfunction of The Pacing Lead (Product Issues) | 7 (7)
LV Lead Stylet Malfunction (Product Issues) | 1 (1)
Oversensing (Product Issues) | 1 (1)
Pectoral/Diaphragmatic/Phrenic Nerve Stimulation (Product Issues) | 104 (124)
Rise in Threshold and Exit Block (Product Issues) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT02832622/Prot_SAP_000.pdf